CLINICAL TRIAL: NCT04146324
Title: A Prospective Observational Study in Patients Receiving Adjuvant Nivolumab Therapy for Resected Melanoma in Australia
Brief Title: An Observational Study of Adjuvant (Post-surgery) Therapy With Nivolumab for Resected (Completely Removed) Melanoma in Australia
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-7CK
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Melanoma
Keywords: Adjuvant; nivolumab
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adjuvant nivolumab therapy: Participants receiving nivolumab as an adjuvant therapy according to the market authorization in Australia
  Interventions: Drug: nivolumab

INTERVENTIONS:
Drug: nivolumab — Administered as adjuvant therapy as per the market authorization in Australia

SUMMARY:
This study is designed to estimate the effectiveness of nivolumab when given to participants after removing their cancer with surgery, over a 5-year follow-up, in real-world conditions in Australia.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Adults with a primary diagnosis of melanoma with involvement of lymph nodes or metastatic disease who have undergone complete surgical removal and have no evidence of disease
* Decision to treat with adjuvant nivolumab therapy has already been taken
* Ability to provide written informed consent to participate in the study

Exclusion Criteria:

* Adults with a current diagnosis of persisting advanced melanoma
* Adults currently enrolled in an interventional clinical trial for his/her melanoma treatment

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults whose melanoma had spread to the lymph nodes or other parts of the body and was surgically removed, and who are receiving post-surgery treatment with nivolumab to decrease the risk of cancer coming back.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Relapse-Free Survival (RFS) | Up to 5 years post treatment initiation with adjuvant nivolumab therapy
  The time between the date of randomisation and the date of first recurrence, new primary melanoma, or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Percentage of Participants with Distant Metastasis-Free Survival (DMFS) | Up to 5 years post treatment initiation with adjuvant nivolumab therapy
Overall Survival (OS) | Up to 5 years post treatment initiation with adjuvant nivolumab therapy
Description of sociodemographic profile of participants | At treatment initiation with adjuvant nivolumab therapy
Description of clinical characteristics of participants | At treatment initiation with adjuvant nivolumab therapy
Prior medical history of participants | At treatment initiation with adjuvant nivolumab therapy
Description of nivolumab pattern of use | At treatment initiation with adjuvant nivolumab therapy
Health-related quality of life (HRQOL) of participants as assessed by European Quality of Life Five Dimensional Scale (EuroQOL-5D/EQ-5D) | Up to 5 years post treatment initiation with adjuvant nivolumab therapy
HRQOL of participants as assessed by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ C-30) | Up to 5 years post treatment initiation with adjuvant nivolumab therapy
HRQOL of participants as assessed by Functional Assessment of Cancer Therapy-Melanoma (FACT-M) questionnaire | Up to 5 years post treatment initiation with adjuvant nivolumab therapy
Participants' socioeconomic status as assessed by their highest education level | At treatment initiation with adjuvant nivolumab therapy
Description of care received as assessed by Healthcare Resource Utlization | During, and up to 5 years post discontinuation of nivolumab use
Number of participants experiencing immune-related Adverse Events (AEs) | Up to 5 years post treatment initiation with adjuvant nivolumab therapy
Number of participants experiencing non-immune-related AEs | Up to 5 years post treatment initiation with adjuvant nivolumab therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- Australia (9):
  - Local Institution, Garran, Australian Capital Territory
  - Local Institution, Birtinya, Queensland
  - Local Institution, Cairns, Queensland
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Herston, Queensland
  - Local Institution, Woolloongabba, Queensland
  - Local Institution - 0006, Woodville South, South Australia
  - Local Institution, Box Hill, Victoria
  - Local Institution, Malvern, Victoria

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm